CLINICAL TRIAL: NCT05655468
Title: Effect of Prolonged Use of Dronedarone on Recurrence in Patients With Non-paroxysmal Atrial Fibrillation After Radiofrequency Ablation
Acronym: DORIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Yang Bing, deputy director of cardiovascular department, Shanghai East Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFLC2022011
Record Dates: First submitted 2022-12-07; First posted 2022-12-19 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
Keywords: dronedarone; placebo; non-paroxysmal atrial fibrillation; ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dronedarone (Experimental): dronedarone 400mg twice a day for 9 months
  Interventions: Drug: Dronedarone
- placebo (Placebo Comparator): Placebo(for dronedarone ) a day for 9 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronedarone — oral administration fed conditions
  Arms: dronedarone
Drug: Placebo — strictly identical in appearance with dronedarone,oral administration fed conditions
  Arms: placebo

SUMMARY:
Recurrence rate remains high after radiofrequency ablation in patients with non-paroxysmal atrial fibrillation(AF). Prolonged use of anti-arrhythmic drugs (AAD) beyond the post-ablation blanking has been adopted as a solution but without sufficient clinical evidence. Dronedarone is an AAD valid to maintain sinus rhythm and has fewer side effect than other AAD for long-term use.We sought to investigate the effect of prolonged use of dronedarone on recurrence of non-paroxysmal AF patients beyond the post-blanking period within the first year after ablation.

DETAILED DESCRIPTION:
In this multicenter, randomized, placebo-controlled trial, patients with non-paroxysmal AF will receive dronedarone for three months after radiofrequency ablation. Eligible Patients will then be randomly divided into dronedarone and placebo groups and followed up until one year after ablation. The primary endpoint is the cumulative nonrecurrence rate post three months and within one year after ablation. 7-day Holter monitoring (ECG patch) will be scheduled at 6,9, and 12 months after ablation for evaluating AA recurrence. Secondary endpoints include dronedarone withdrawal due to side effect or intolerance of AA recurrence, time to the first recurrence, repeat ablation, electrical cardioversion, unscheduled visit ,and rehospitalization.

This trial will evaluate whether prolonged use of dronedarone effectively reduces recurrence rate after ablation in non-paroxysmal AF patients. The result of this trial will provide evidence for optimizing post-ablation anti-arrhythmic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years;
2. Diagnosis of non-paroxysmal AF
3. Undergoing AF ablation for the first time

Exclusion Criteria:

1. Unwilling to take or intolerant to dronedarone;
2. Hypersensitivity to the drug ingredient
3. Patients with decompensated heart failure, class NYHA IV, or left ventricular ejection fraction (LVEF) ≤40%
4. Bradycardia <50 bpm
5. QTc Bazett interval ≥500ms or PR interval >280ms
6. II or III atrioventricular (AV) block or sick-sinus syndrome without permanent pacemaker
7. Diagnosed with acute coronary syndrome or treated with percutaneous coronary intervention within the last 3 months
8. Patients with structural heart disease (moderate to severe aortic or mitral valve stenosis, interventricular septal thickness >15mm, congenital heart disease)
9. Accepted cardiac surgery within the last 3 months
10. Left atrial diameter (LAD) >55 mm
11. Patients with left atrial or left auricular thrombosis
12. Patients with Hyperthyroidism
13. Severe dysfunction of liver and kidney diseases (ALT≥3ULN or eGFR<30ml/min/1.73m2)
14. Abnormal blood coagulation
15. Concomitant use of dabigatran
16. Concomitant use of drugs that prolong QTc or may induce torsades de pointes
17. Concomitant use of strong CYP3A inhibitors
18. Concomitant use of another Class IA, IC, or III AADs
19. Patients suffering from serious infection, mental illness or malignant tumors
20. Pregnancy or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
cumulative nonrecurrence rate | post 3 to 12 months after ablation
  defined as any atrial tachyarrhythmias (including atrial fibrillation, atrial flutter, or atrial tachycardia) recorded by electrocardiogram (ECG)>30s

SECONDARY OUTCOMES:
drug withdrawal because of side effect | post 3 to 12 months after ablation
drug withdrawal due to intolerance to or persistent AA(lasting more than 7 days) | post 3 to 12 months after ablation
time to first recurrence | post 3 to 12 months after ablation
cardioversion due to recurrence | post 3 to 12 months after ablation
repeat ablation due to recurrence | post 3 to 12 months after ablation
unscheduled visit and rehospitalization due to recurrence | post 3 to 12 months after ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

REFERENCES:
- [Derived] Wu Y, Fan F, Yu J, Zhou J, Xie X, Xia G, Zhong D, Cheng D, Zhang B, Wang X, Chen Z, Wang S, Li X, Yang B. Effect of Prolonged Use of Dronedarone on Recurrence in Patients with Non-Paroxysmal Atrial Fibrillation After Radiofrequency Ablation (DORIS): Rationale and Design of a Randomized Multicenter, Double-Blinded Placebo-Controlled Trial. Cardiovasc Drugs Ther. 2024 Oct;38(5):1047-1052. doi: 10.1007/s10557-023-07460-1. Epub 2023 May 8. PMID 37155004